CLINICAL TRIAL: NCT05221827
Title: Clinical Performance Evaluation of the C2i-Test for Detecting Molecular Residual Disease (MRD) in Bladder Cancer Patients.
Brief Title: Clinical Performance Evaluation of the C2i-Test
Status: Terminated | Type: Observational
Why Stopped: Not in line with company's recently updated clinical development strategy
Sponsor: C2i Genomics (Industry)
Collaborators: New Jersey Urology (Unknown); University of Texas (Other); Baylor College of Medicine (Other); NY Health d/b/a New York Cancer and Blood Specialists (Other); The Cleveland Clinic (Other); Fox Chase Cancer Center (Other); New York University (Other); University of Washington (Other); Oregon Health and Science University (Other); University of Southern California (Other); Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: CA-F01-02
Record Dates: First submitted 2022-01-19; First posted 2022-02-03 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Muscle-Invasive Bladder Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MIBC: Patients with clinically and pathologically confirmed diagnosis of MIBC stage II-IIIA, planned to undergo RC.
  Interventions: Diagnostic Test: C2i Test

INTERVENTIONS:
Diagnostic Test: C2i Test — The C2i-Test, a personalized molecular circulating tumor DNA (ctDNA) test, is an in vitro qualitative test that uses next generation sequencing (NGS)-based whole-genome sequencing (WGS) data for detecting molecular residual disease (MRD).

SUMMARY:
The C2i-WGS-MRD Test (hereinafter referred to as C2i-Test), a personalized molecular circulating tumor DNA (ctDNA) test, is an in vitro qualitative test that uses next generation sequencing (NGS) based whole-genome sequencing (WGS) data for detecting molecular residual disease (MRD) in patients diagnosed with muscle-invasive bladder cancer (MIBC) and histopathologically classified as stage II-IIIA. The C2i-Test is a single site assay performed in the C2i Genomics' CLIA-certified laboratory. This is a prospective non-interventional study to collect definitive evidence of the safety and effectiveness of C2i-Test for the intended use, in a statistically justified number of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have clinically and pathologically confirmed diagnosis of MIBC.
* A representative FFPE biopsy specimen (from the transurethral resection of bladder tumor - TURBT) with at least 1 H&E slide and 9 unstained slides, with an associated pathology report must be available.
* Subjects must agree to 8mL blood collection during all visits.
* Participants with MIBC, clinical stage II (cT2, N0) or IIIA (cT3, N0; cT4a, N0; cT1-T4a, N1) (lymph node positive if >10 mm on CT or MRI in short axis), diagnosed by work-up recommended by NCCN guidelines (including cystoscopy, abdominal/pelvic imaging that includes imaging of upper urinary tract collecting system, examination under anesthesia, TURBT, and bone imaging if clinical suspicion or symptoms of bone metastases within 4 weeks prior to enrollment, however patients can be enrolled if they are reassessed, and the localized status is reconfirmed with subsequent imaging studies).
* Histopathologically confirmed urothelial carcinoma as diagnosed by TURBT. Variant urothelial histology (e.g., micropapillary, plasmacytoid, sarcomatoid, nested variant, lymphoepithelioid, nested variant) is acceptable. Mixed histology (adenocarcinoma, squamous cell) is acceptable if there is a predominant (>50%) urothelial component.
* Treatment plans must include RC.
* Participant is willing and able to comply with the protocol, including RC, pelvic lymph node dissection (PLND), and prostatectomy (if applicable).
* The patient must be deemed appropriate for RC, PLND, and prostatectomy (if applicable) by his/her oncologist and/or urologist.
* Patient's treatment plan may or may not include neoadjuvant treatment and/or adjuvant treatment.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
* Patient is willing and able to provide written informed consent for samples to be collected and used in this study.

Exclusion Criteria:

* Extravesical urothelial carcinoma (UC) that invades the pelvic and/or abdominal wall for bladder cancer (T4b) as evidenced by imaging.
* Evidence of UC in the urinary tract (ureters, renal pelvis, and urethra) as evidenced by work-up in accordance with NCCN guidelines (e.g., abdominal/pelvic imaging) that includes imaging of upper urinary tract collecting system).
* Clinical evidence of greater than 1 positive LN (≥ 10 mm in short axis) or metastatic bladder cancer per IV contrast-enhanced CT or MRI scan and/or PET-CT scan.
* Patients with mixed histology and <50% urothelial component as evidenced by TURBT pathology.
* Tumors that contain any neuroendocrine/small cell component as evidenced by TURBT pathology.
* Diagnosis of 3 or more synchronous cancers.
* Malignancies other than urothelial cancer within 5 years prior to study entry except those with negligible risk of metastases or death and treated with the expectation of curative outcome (such as: carcinoma in situ of the cervix, basal or squamous cell skin cancer, ductal carcinoma in situ treated surgically with curative intent, papillary thyroid carcinoma, localized prostate cancer treated with curative intent and absence of prostate-specific antigen (PSA) relapse, or incidental prostate cancer [Gleason score ≤ 3 + 4 and PSA < 10 ng/mL] undergoing active surveillance and treatment naïve).
* Prior chemotherapy or immunotherapy, radiation therapy, or surgery other than TURBT for bladder cancer.
* Per physician discretion: patients with severe or uncontrolled concomitant medical, surgical, or psychiatric disease that could affect compliance with the protocol, the results of the study, or interpretation of the results.
* Individuals who cannot provide consent for their own participation will not be included.
* Sponsors employees and their family.

Ages: 22 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with clinically and pathologically confirmed diagnosis of MIBC stage II-IIIA, planned to undergo RC.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Overall specificity of the C2i-Test | 3-year
  Predicting 3-year recurrence-free survival post- definitive treatment (RC/RC + adjuvant chemotherapy), compared to the GS diagnosis as determined by patient outcome (based on NCCN guidelines).

SECONDARY OUTCOMES:
Overall sensitivity of the C2i-Test | 3-year
  Predicting non-pCR following neoadjuvant treatment completion prior to RC, compared to the GS diagnosis as determined by the pathology report.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Lotan, MD, Principal Investigator — UT Southwestern
Locations (1):
- New Jersey Urology, Bloomfield, New Jersey, United States